CLINICAL TRIAL: NCT07318974
Title: Preliminary Assessment of the Impact of Melatonin Therapy for Women With Diminished Ovarian Reserve on the Ovarian Reserve and the ICSI Outcomes
Brief Title: Melatonin Therapy for Improving ICSI Outcomes in Women With Diminished Ovarian Reserve
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Basma Sakr, Professor of Obstetrics & Gynecology, Faculty of Medicine, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rc 2.8.2025
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: ICS
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin Group (Active Comparator): Participants receive one 3 mg Melatonin capsule orally every night for 28 consecutive days prior to the start of ovarian stimulation for ICSI.
  Interventions: Drug: Melatonin capsule
- Placebo Group (Active Comparator): Participants receive an identical-appearing placebo capsule orally every night for 28 consecutive days prior to the start of ovarian stimulation for ICSI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin capsule — Participants receive 3mg of Melatonin Capsules
  Dosage & Frequency: Once at night
  Duration: The treatment continues for 28 days
  Arms: Melatonin Group
Drug: Placebo — Participants receive identical-appearing placebo capsule
  Dosage & Frequency: Once at night
  Duration: The treatment continues for 28 days
  Arms: Placebo Group

SUMMARY:
Diminished ovarian reserve (DOR) is a major challenge in female fertility, often leading to poor oocyte quality and low pregnancy rates during assisted reproduction. Melatonin is a potent antioxidant that may protect developing eggs from oxidative stress. This randomized clinical trial aims to evaluate whether a 4-week course of oral melatonin therapy before egg retrieval can improve the quality of oocytes and embryos, and ultimately increase pregnancy rates for women with DOR undergoing Intracytoplasmic Sperm Injection (ICSI). The study compares melatonin therapy against a placebo to assess its impact on follicular fluid health and clinical pregnancy success.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diminished Ovarian Reserve (DOR) based on Bologna criteria (e.g., low AMH, low AFC).
* Undergoing ICSI with frozen blastocyst transfer (FBT) protocol.
* Willingness to comply with a 28-day pre-retrieval medication regimen.

Exclusion Criteria:

* Severe endometriosis or hydrosalpinx.
* Uterine anomalies (e.g., large fibroids or uterine septums).
* Chronic systemic diseases (e.g., uncontrolled diabetes or hypertension).
* Partner with severe male factor infertility requiring TESE/PESA (to isolate the effect on oocyte quality).
* Current use of other antioxidant supplements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The Success Rate of Treatment Regimens in Achieving Clinical Pregnancy | 2-3 Months
  The proportion of patients who achieved a clinical pregnancy (confirmed by ultrasound visualization of a gestational sac with fetal heart activity) following frozen blastocyst transfer, reflecting the effectiveness of the administered melatonin therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El Qalyoubia, Egypt